CLINICAL TRIAL: NCT06162702
Title: To Investigate the Efficacy and Safety of Fecal Microbiota Transplantation (FMT) in the Treatment of Small Intestinal Bacterial Overgrowth (SIBO).
Brief Title: Clinical Study of Fecal Microbiota Transplantation in the Treatment of Small Intestinal Bacterial Overgrowth (SIBO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMT-SIBO
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Small Intestinal Bacterial Overgrowth; Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT Responder (Experimental)
  Interventions: Procedure: Fecal microbiota transplantation
- FMT non-Responder (Experimental)
  Interventions: Procedure: Fecal microbiota transplantation

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — Fecal microbiota transplantation (FMT) achieves the purpose of treating intestinal and extra-intestinal diseases by transplanting the functional microbes in the feces of healthy people into the patient's intestine through the upper or lower alimentary tract routes to rebuild the patient's intestinal microbiota.

SUMMARY:
Small intestinal bacterial overgrowth (SIBO) is defined as the presence of excessive numbers of bacteria in the small bowel causing gastrointestinal (GI) symptoms. These bacteria are usually coliforms, which are typically found in the colon and include predominantly Gram-negative aerobic and anaerobic species that ferment carbohydrates producing gas .Fecal Microbiota Transplantation (FMT) is a therapeutic method to transplant the microbiota from the feces of healthy people into the intestinal tract of patients. To explore the overall efficacy and safety of FMT in the treatment of SIBO.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a positive breath test result upon initial admission.
* Patients presenting with abdominal symptoms.
* Patients who have stool and small intestinal fluid samples available before and after FMT.

Exclusion Criteria:

* Patients with gastrointestinal malignancies.
* Patients with a history of gastrointestinal surgery.
* Patients on long-term probiotic use.
* Patients with a history of extensive antibiotic use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (Assessing the safety of FMT in patients with SIBO) | 7 days, 1 month
  Document adverse events related to FMT that occurred during the study, including their frequency and severity.
Number of Patients with gastrointestinal symptom scores | 7 days, 1 month
  The efficacy of FMT in SIBO patients was evaluated according to the scores of gastrointestinal symptoms before and after treatment. Patients with gastrointestinal symptom scores, including some of the abdominal symptoms and defecation situation, we can according to this questionnaire to assess patients with abdominal symptoms and defecate on the improvement of their situation.
Investigating the impact of FMT on the colonic and small intestinal microbiota. | 7 days, 1 month
  For patients before and after the FMT feces and small intestinal juice samples 16 s rRNA sequencing, compare the difference between before and after the FMT feces and bacteria in the intestinal flora of diversity, species composition belong. The changes of commensal bacteria, opportunistic pathogens and pathogenic bacteria in feces and small intestinal fluid after FMT were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Intestinal Microenvironment Treatment Center of General Surgery, Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No